CLINICAL TRIAL: NCT04829786
Title: A Double-Blind, Randomized, Cross-Over Single-Dose Study to Compare the Pharmacokinetics, Safety, and Tolerability Following Administration of Palovarotene in Healthy Japanese and Non-Asian Subjects
Brief Title: Study to Compare the Pharmacokinetics, Safety, and Tolerability Following Administration of Palovarotene in Healthy Japanese and Non-Asian Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Clementia Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Organization: Ipsen (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PVO-1A-101
Record Dates: First submitted 2021-04-01; First posted 2021-04-02 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-04

CONDITIONS: FOP
MeSH Terms: interventions — Palovarotene

STUDY DESIGN:
Intervention Model Description: The subjects will be randomized to receive in Period 1 either the low-dose or high-dose first, and in Period 2 they received the alternate dose.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Japanese group (Experimental): The subjects will receive in Period 1 either the low-dose or high-dose first, and in Period 2 they will receive the alternate dose. There is a washout period between periods.
  Interventions: Drug: palovarotene low-dose; Drug: palovarotene high-dose
- non-Asian group (Experimental): The subjects will receive in Period 1 either the low-dose or high-dose first, and in Period 2 they will receive the alternate dose. There is a washout period between periods.
  Interventions: Drug: palovarotene low-dose; Drug: palovarotene high-dose

INTERVENTIONS:
Drug: palovarotene low-dose — oral capsules
Drug: palovarotene high-dose — oral capsules

SUMMARY:
this study purpose is to assess safety, tolerability and the pharmacokinetic (PK) profile of palovarotene in healthy Japanese and matched (with respect to sex, age, and weight) non-Asian subjects aged 18 to 55 years.

ELIGIBILITY:
Key Inclusion Criteria:

* The subject had a body mass index (BMI) of 18 to 30 kg/m2 and a body weight of 50 kg or more. Body mass index was calculated as follows: weight (kg)/height2 (m2).
* The subject had a resting (at least 5 minutes) sitting pulse of greater than 45 but less than 100 beats per minute (BPM) and systolic and diastolic blood pressure (BP) of less than 140/90 mmHg
* The subject was a nonsmoker for at least 6 months prior to the screening visit and had a maximum smoking history of 5-pack years
* The subject was in good general health as determined by medical history, physical examination, 12-lead ECG, vital signs, and clinical laboratory results obtained within 28 days prior to the start of the study.
* The subject had the ability to swallow an oral solid-dosage form of medication

Non-Asian Subjects:

* The subject must have had both biological parents and four biological grandparents of non-Asian descent.
* The subject must have been matched individually (on a 1:1 basis) with respect to sex, age (within 5 years), and weight (within 10%) to a Japanese subject.

Japanese Subjects

* The subject must have been born in Japan and have both biological parents and four biological grandparents of Japanese descent.
* The subject had a valid Japanese passport.
* The subject must have lived outside of Japan for no more than 5 years.
* The subject must not have significantly changed their diet since leaving Japan, eg, he/she must mainly had been eating a "Japanese" diet.

Key Exclusion Criteria:

* The subject had a history or current evidence of a clinically significant or uncontrolled disease, including but not limited to: cardiovascular, hepatic, renal, hematological, neuropsychological, endocrine, gastrointestinal, reproductive, or pulmonary.
* The subject was pregnant, nursing, or planned to become pregnant or donate gametes (ova or sperm) for in vitro fertilization during the study period or for 30 days following the subject's last study-related visit (for eligible subjects only, if applicable).
* The subject had a medical condition that may have potentially been aggravated by a systemic retinoid such as isotretinoin or etretinate.
* The subject had been exposed to synthetic oral retinoids in the past 30 days prior to the screening visit (signature of the informed consent).
* The subject was currently using vitamin A or beta carotene, multivitamins containing vitamin A or beta carotene, or herbal preparations, fish oil, and was unable or unwilling to discontinue use of these products for the duration of the study.
* The subject had a history or presence of silent infections, including positive tests for human immunodeficiency virus type 1 (HIV-1), HIV-2, hepatitis B virus (HBV), or hepatitis C virus (HCV).
* The subject had any disease or condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
* The subject had concurrent treatment with tetracycline due to the potential increased risk of pseudotumor cerebri.
* The subject had a history of allergy or hypersensitivity to retinoids or lactose.
* The subject had been exposed to any investigational drug within 30 days or six half-lives (whichever is greater) of the screening visit.
* The subject had been treated with any known CYP450 3A4 inhibitors (eg, ketoconazole, gestodene, rifampin) within 30 days prior to the screening visit.
* The subject had a history of alcohol and/or substance abuse.
* The subject was considered to be vulnerable (eg, cognitively impaired, a person kept in detention).
* Any reason that in the opinion of the Investigator would have led to the inability of the subject and/or family to comply with the protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2015-10-23 (Actual); Study Completion 2015-10-23 (Actual)

PRIMARY OUTCOMES:
Maximum (peak) plasma drug concentration | pre-dose (0 hour), 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, and 72 hours post-drug administration.
Time to reach maximum (peak) plasma concentration following drug administration | pre-dose (0 hour), 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, and 72 hours post-drug administration.
Area under the plasma concentration time curve from time zero to the last quantifiable time point, calculated by linear-log trapezoidal summation | pre-dose (0 hour), 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, and 72 hours post-drug administration.
Area under the plasma concentration time curve from time zero to infinity, calculated by linear-log trapezoidal summation and extrapolated to infinity by addition of the last quantifiable plasma concentration divided by the elimination rate constant | pre-dose (0 hour), 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, and 72 hours post-drug administration.
Terminal disposition rate constant/terminal rate constant, determined by linear regression of the terminal points of the log-linear plasma concentration-time curve | pre-dose (0 hour), 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, and 72 hours post-drug administration.
Elimination half-life | pre-dose (0 hour), 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, and 72 hours post-drug administration.
Apparent volume of distribution after non-intravenous (oral) administration | pre-dose (0 hour), 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, and 72 hours post-drug administration.
Apparent total clearance of the drug from plasma after oral administration calculated by dose/ AUC(0-∞) | pre-dose (0 hour), 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, and 72 hours post-drug administration.

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen